CLINICAL TRIAL: NCT00383344
Title: Phase II Study on the Role of the Positron Emission Tomography Combined With CT Scan for the Evaluation on Crohn Disease
Brief Title: Use of FDG PET/CT to Evaluate Crohn Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eric Turcotte (Other)
Responsible Party: Sponsor-Investigator, Eric Turcotte, MD, Université de Sherbrooke
Organization: Université de Sherbrooke (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 06-086
Record Dates: First submitted 2006-10-02; First posted 2006-10-03 (Estimated); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Crohn Disease
Keywords: Crohn Disease; Positron Emission Tomography; Colonoscopy
MeSH Terms: conditions — Crohn Disease

INTERVENTIONS:
Procedure: FDG PET/CT

SUMMARY:
The purpose of this study will permit to determine the role of FDG PET/CT to diagnose Crohn Disease and recurrence of Crohn disease after having compared results of PET/CT's with results of exams routinely performed(colonoscopy and bowel follow through).

DETAILED DESCRIPTION:
Crohn disease is an inflammatory disease of the digestive system that may affect the small and large intestines. Remission and recurrence clinically characterized its development. When recurrence occurs, a careful examination is necessary in order to determine the extent and the severity of the disease. Actual exams performed are invasive and uncomfortable(colonoscopy and bowel follow through). Compare to these exams, PET/CT is less fierce to undergo and has less risks. Two groups are proposed in this project: 15 patients will be enroll in the active disease group and 15 patients will be enroll in the remission group. In regards of the area and the extent of the disease,PET/CT exams shall provide similar information than what usual tests provide. PET/CT exams shall also provide more information in order to better differentiate inflammatory stenosis from scars stenosis especially located in the small intestine.

ELIGIBILITY:
Inclusion Criteria:

* Men or women known having a Crohn's disease de novo diagnosis or a Crohn's disease recurrence based on a seven days questionnaire and a physical exam.
* Men or women with a past history of Crohn's disease but considered clinically in remission based on a seven days questionnaire, a physical exam and a Crohn's disease activity index (CDAI) score < to 150.

Exclusion Criteria:

* Men or women less than 18 years of age
* Pregnancy
* Breastfeeding
* Renal failure
* Suspicion of a Crohn's disease infectious complication (abscess,fistula)
* Infectious colitis determined at the initial checkup
* Diabetes
* Severe allergy to iode contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-10-01 (Actual); Primary Completion 2007-05-01 (Actual); Study Completion 2007-05-01 (Actual)

PRIMARY OUTCOMES:
Diagnosis of Crohn Disease de novo and Crohn Disease recurrences with FDG PET/CT.

SECONDARY OUTCOMES:
Detection of inflammatory areas not suspected with usual tests
Detection of an inflammatory activity for remission patients

CONTACTS AND LOCATIONS:
Overall Officials: François Bénard, MD, Principal Investigator — Université de Sherbrooke
Locations (1):
- CHUS/CRC, Sherbrooke, Quebec, Canada